CLINICAL TRIAL: NCT05881109
Title: Population Pharmacokinetics and Dose Optimization of Caspofungin in Adolescents With Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Population Pharmacokinetics and Dose Optimization of Caspofungin in Adolescents
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, professor, Shandong University
Other Study IDs: caspofungin-001
Record Dates: First submitted 2023-05-12; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Invasive Fungal Infections
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Caspogunfin — No specific interventions were administrated. Participants receive interventions as part of routine medical care, where CAS was infused intravenously over 60 min at a loading dose of 70 mg/m2 on day 1, followed by a maintenance dose of 50 mg/m2 (maximum: 70 mg daily).

SUMMARY:
Caspofungin (CAS) is used to prevent and treat invasive fungal infections patients older than 3 months. However, the optimal dosing strategy of CAS is lacking in adolescents from 12 to 17 years old, especially those undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT), who are vulnertable to fungal infections. The study aimed to establish a population pharmacokinetic (PPK) model and assess the dosing schemes of CAS in adolescents with allogeneic hematopoietic stem cell transplantation (allo-HSCT).

ELIGIBILITY:
Inclusion Criteria:

* The adolescents (12 - 17 years) underwent allo-HSCT
* Use caspofungin for the prevention or treatment of fungal infections

Exclusion Criteria:

* Intolerable to caspofungin
* Participate into other clinical studies
* There are conditions that researchers do not consider it appropriate to join the research.

Ages: 12 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: The adolescents (12 - 17 years old) undergoing allo-HSCT and receiving CAS as prevention or treatment for IFIs
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
The PTAs of AUC24/MIC90 for C. albicans , C. glabrata , and C. parapsilosis | 1 day
  The probability of target attainment (PTA) of the ratio of AUC24 (area under the concentration-time curve from 0 to 24 hours) and MIC90 (the lowest concentration of caspofungin at which 90% of the isolates were inhibited) (AUC24/MIC90) for C. albicans (0.06 mg/L), C. glabrata (450 mg/L), and C. parapsilosis (1185 mg/L) .
The PTAs of AUC24/MIC for various species of Candida spp isolates | 1 day
  The probability of target attainment (PTA) of the ratio of AUC24 (area under the concentration-time curve from 0 to 24 hours) and MIC (minimal inhibitory concentration) (AUC24/MIC) for various species of Candida spp isolates with a MIC range of 0.03 to 1.0 mg/L
The PTAs of trough concentration | the trough concentration (24 hours after administration) at the steady state
  PTA of patients with CAS trough concentration ≥ 1 μg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Children's Hospital, Wuhan, China